CLINICAL TRIAL: NCT01904643
Title: A Phase I Study of Lenalidomide Therapy Prior to Re-induction Chemotherapy With Mitoxantrone, Etoposide, and Cytarabine (MEC) for the Treatment of Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: Lenalidomide and Combination Chemotherapy in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Accrual factor
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Iberri, Clinical Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-27313; NCI-2013-01349 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB-27313 (Other: Stanford IRB); P30CA124435 (NIH); HEMAML0024 (Other: OnCore ID)
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Lenalidomide; Mitoxantrone; Etoposide; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (lenalidomide, combination chemotherapy) (Experimental): LENALIDOMIDE PRIMING: Patients receive lenalidomide PO for 5 or 7 days.
  RE-INDUCTION CHEMOTHERAPY: Patients receive etoposide IV over 1 hour, cytarabine IV over 3 hours, and mitoxantrone hydrochloride IV over 15-30 minutes on days 1-5. Patients failing to achieve blast count < 5% at 21 days may receive a second course of induction therapy. Patients achieving complete remission proceed to lenalidomide priming.
  LENALIDOMIDE PRIMING: Within 4-6 weeks, patients receive lenalidomide PO for 5 or 7 days and then proceed to consolidation therapy.
  CONSOLIDATION CHEMOTHERAPY: Patients receive etoposide IV over 1 hour, cytarabine IV over 3 hours, and mitoxantrone hydrochloride IV over 15-30 minutes on days 1-4. Treatment repeats every 28-35 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lenalidomide; Drug: mitoxantrone hydrochloride; Drug: etoposide; Drug: cytarabine

INTERVENTIONS:
Drug: lenalidomide — Given PO
  Other Names: CC-5013; IMiD-1; Revlimid
Drug: mitoxantrone hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Novantrone
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside

SUMMARY:
This phase I trial studies the side effects and the best dose of lenalidomide when given together with combination chemotherapy in treating patients with relapsed or refractory acute myeloid leukemia. Lenalidomide may stop the growth of acute myeloid leukemia by blocking blood flow to the cancer. Drugs used in chemotherapy, such as mitoxantrone hydrochloride, etoposide, and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving lenalidomide and combination chemotherapy may be an effective treatment for acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of lenalidomide when used in combination with mitoxantrone hydrochloride, etoposide, and cytarabine (MEC) in patients with relapsed or refractory acute myeloid leukemia (AML).

II. To determine the dose-limiting toxicities (DLTs) of this combination in this patient population.

SECONDARY OBJECTIVES:

I. To determine whether the combination of lenalidomide priming prior to re-induction chemotherapy with MEC has clinical activity in patients with relapsed or refractory AML.

OUTLINE: This is a dose-escalation study of lenalidomide.

LENALIDOMIDE PRIMING: Patients receive lenalidomide orally (PO) for 5 or 7 days.

RE-INDUCTION CHEMOTHERAPY: Patients receive etoposide intravenously (IV) over 1 hour, cytarabine IV over 3 hours, and mitoxantrone hydrochloride IV over 15-30 minutes on days 1-5. Patients failing to achieve blast count < 5% at 21 days may receive a second course of induction therapy. Patients achieving complete remission proceed to lenalidomide priming.

LENALIDOMIDE PRIMING: Within 4-6 weeks, patients receive lenalidomide PO for 5 or 7 days and then proceed to consolidation therapy.

CONSOLIDATION CHEMOTHERAPY: Patients receive etoposide IV over 1 hour, cytarabine IV over 3 hours, and mitoxantrone hydrochloride IV over 15-30 minutes on days 1-4. Treatment repeats every 28-35 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible include those with diagnosis of AML other than acute promyelocytic leukemia by World Health Organization (WHO) criteria with relapsed disease after induction therapy or refractory to induction chemotherapy, as determined by morphology on bone marrow biopsy; also eligible are patients unwilling to receive standard induction chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Serum creatinine =< 1.5 mg/dL; if serum creatinine > 1.5 mg/dL, then the estimated glomerular filtrate rate (GFR) must be > 60ml/min/1.73m^2 as calculated by the Modification of Diet in Renal Disease equation
* Serum bilirubin =< 1.5 x upper limit of normal (ULN) unless elevation is considered to be secondary to Gilbert's syndrome, hemolysis, or hepatic infiltration by AML
* Aspartate transaminase (AST)/alanine transaminase (ALT) =< 2.5 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* All study participants must be registered into the mandatory Revlimid assistance (RevAssist) program, and be willing and able to comply with the requirements of RevAssist
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for cycle 1 (prescriptions must be filled within 7 days as required by RevAssist) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy

Exclusion Criteria:

* Patient must not undergo concomitant radiotherapy, chemotherapy or immunotherapy; patient must not be in concurrent study with other investigational agents
* Patients who have received prior lenalidomide therapy are not eligible for this study; further there should be at least a 14-day window from the patient's last prior therapy before initiation of treatment on clinical trial
* Have other severe concurrent disease or serious organ dysfunction involving the heart, kidney, liver or other organ system that may place the patient at undue risk to undergo treatment
* Have significant, uncontrolled active infection
* Pregnant or nursing patients will be excluded from the study
* Known human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05-13 (Actual); Study Completion 2015-07-18 (Actual)

PRIMARY OUTCOMES:
MTD of lenalidomide when used in combination with MEC determined by DLT using the Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 | 42 days
  Hematologic and non-hematologic toxicities will be tabulated.

SECONDARY OUTCOMES:
Response rate (complete remission [CR], CR with incomplete blood count recovery [CRi], partial remission [PR] or stable disease [SD]) using LeukemiaNet guidelines | Up to 6 months
  Proportions of these patients in each response category will be tabulated; the combined proportion in categories CR, CRi, PR, and SD will be computed along with an exact 95% confidence interval.
Response duration | From start of induction, assessed up to 6 months
  Summarized using a Kaplan-Meier plot.
Early mortality | From start of induction, assessed up to 6 months
  Summarized using a Kaplan-Meier plot.

CONTACTS AND LOCATIONS:
Overall Officials: David Iberri, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No